CLINICAL TRIAL: NCT01850654
Title: Ohio Colorectal Cancer Prevention Initiative: Universal Screening for Lynch Syndrome
Brief Title: Ohio Colorectal Cancer Prevention Initiative
Acronym: OCCPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Heather Hampel, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-12170
Record Dates: First submitted 2013-05-03; First posted 2013-05-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Lynch Syndrome; Colorectal Cancer
Keywords: colorectal cancer; colon cancer; rectal cancer; endometrial cancer; Lynch syndrome; Ohio colon cancer study; OSU colon study
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Endometrial Neoplasms | interventions — Methylation; Genetic Testing; Genetic Counseling; Biological Specimen Banks; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probands (Other): Participants with colorectal or endometrial cancer.
  Interventions: Genetic: LS tumor screening; Genetic: Genetic testing; Behavioral: Genetic Counseling; Other: Biorepository; Behavioral: Questionnaire
- First-degree relatives of the participants with CRC (Other): The first-degree relatives of the CRC probands (participants with colorectal cancer).
  Interventions: Other: Biorepository; Behavioral: Questionnaire
- At-risk relatives (Other): The relatives of the participants found to have Lynch syndrome.
  Interventions: Genetic: Genetic testing; Behavioral: Genetic Counseling; Other: Biorepository; Behavioral: Questionnaire

INTERVENTIONS:
Genetic: LS tumor screening — All participants with CRC or EC will have LS tumor screening (MSI, IHC, methylation if applicable).
  Other Names: MSI; IHC; Methylation
  Arms: Probands
Genetic: Genetic testing — Next-generation sequencing panel of several genes that increase the risk for hereditary cancers including the LS genes (MLH1, MSH2, MSH6, PMS2, EPCAM), polyposis genes (MUTYH, APC), and others.
  The following study participants will have free genetic testing:
  * CRC and EC study participants with unmethylated MSI-high (MSI-H) tumors
  * CRC and EC study participants with microsatellite stable (MSS) or MSI-low (MSI-L) tumors who have abnormal IHC results and they do not have methylation of the MLH1 promoter
  * CRC study participants diagnosed with CRC <50 years, regardless of tumor studies or family history
  * CRC study participants diagnosed with CRC ≥ 50 years with a FDR with CRC or EC OR synchronous or metachronous CRC or EC throughout their life, regardless of tumor studies.
  At-risk relatives of the individuals found to have LS are eligible for free single site genetic testing.
  Arms: At-risk relatives; Probands
Behavioral: Genetic Counseling — The participants found to have LS or another type of hereditary cancer will have free genetic counseling.
  At-risk relatives of the individuals found to have LS are eligible for free genetic counseling.
  Arms: At-risk relatives; Probands
Other: Biorepository — The biorepository is an optional part of the OCCPI. CRC and EC participants will contribute leftover tumor and blood samples, as well as a saliva sample. FDR of the CRC participants will contribute a saliva sample. The at-risk relatives of those found to have LS will contribute blood and saliva samples.
Behavioral: Questionnaire

SUMMARY:
The purpose of the Ohio Colorectal Cancer Prevention Initiative (OCCPI) is to reduce morbidity and mortality due to colorectal cancer (CRC) in the state of Ohio. By identifying individuals at high-risk for CRC (genetically predisposed) and providing screening recommendations for cancer risk reduction, the OCCPI will understand how to increase length of life and quality of life for those diagnosed with CRC in Ohio, as well as to better prevent CRC in others in Ohio.

Participants will have free tumor screening for Lynch syndrome, and may be eligible for free genetic testing and free genetic counseling as part of this study.

DETAILED DESCRIPTION:
Lynch Syndrome:

Lynch syndrome (LS), previously known as "hereditary non-polyposis colorectal cancer", is a hereditary cancer syndrome that causes the majority of hereditary CRC and approximately 3% of all CRC. LS significantly increases the risk for an individual to develop CRC during their lifetime. Individuals with LS also have an increased risk to develop extracolonic cancers, including endometrial, gastric, ovarian, upper urinary tract, small bowel, biliary tract, CNS, and certain types of skin cancer. Tumor studies, including microsatellite instability (MSI) testing and immunohistochemical (IHC) analysis, provide information regarding characteristic features of LS-associated tumors and can help target genetic testing. Given the hereditary nature of this syndrome, screening all patients who are newly diagnosed with CRC for LS can identify additional individuals who are at high-risk of developing cancer.

Study Aims:

By developing a CRC research infrastructure within the state of Ohio, the OCCPI will achieve the following specific aims:

* Establish and implement a statewide universal screening protocol for LS.
* Elucidate the prevalence of hereditary CRC in Ohio.
* Provide screening recommendations for high-risk individuals with CRC and their families, as well as local access to genetic counseling.
* Create a CRC biorepository for future research on the etiology of CRC from the leftover samples of the CRC patients, as well as samples from their relatives.

With the successful implementation of the OCCPI, knowledge will be gained that will facilitate the adoption of a universal screening protocol for LS in Ohio and the creation of a statewide CRC biorepository to be used for additional studies on cancer risks, prevention, screening, treatment and survivorship.

Study Procedures for CRC and EC participants:

* You will be asked to donate 2-3 tablespoons of blood.
* A small piece of your colorectal or endometrial tumor will be obtained from the hospital where you had your surgery.
* You will be asked to contribute your leftover samples (tumor and blood) to the OCCPI biorepository (sample bank) for help with future research. Additionally, CRC participants will be asked to donate a saliva sample to the OCCPI biorepository. The samples will be kept securely in a lab at OSU. Before your samples can be used for research, the people doing the research must get specific approval from the OCCPI Steering Committee and possibly the Institutional Review Board (IRB) of OSU. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner.
* You will be asked to complete a questionnaire which will ask about your age, medical history, family history, lifestyle factors and environmental exposures. It should take about one hour to complete the questionnaire and you can complete it from home.
* We will test your tumor for features of LS (MSI, IHC, methylation).
* For CRC patients: if your tumor shows features of LS OR you were diagnosed under age 50 OR you have a family history of CRC or endometrial cancer OR you have synchronous or metachronous CRC or endometrial cancer, we will test your blood for the genes that cause LS, as well as other genes that can cause hereditary cancer.
* For endometrial cancer patients: if your tumor shows features of LS, we will test your blood for the genes that cause LS, as well as other genes that can cause hereditary cancer.
* Some patients may have tumor genetic testing.
* If you are found to have LS or another type of hereditary cancer, you will be offered free genetic counseling.
* If you are found to have LS, your at-risk relatives will be offered free genetic counseling and genetic testing.

Study Procedures for first-degree relatives (FDR) of the CRC participants:

The FDRs of all of the CRC study participants will be given the opportunity to contribute to the biorepository for future research.

* Family Member Consent for Contact forms will be provided to the CRC participant at the time of their enrollment for them to distribute to all of their FDRs (parents, siblings and adult children ≥ 25 years). The FDRs will mail the signed form to OSU.
* After obtaining permission to contact the FDRs, OSU will mail them the biorepository consent form and saliva kit to return to the OCCPI biorepository.
* The FDRs of the CRC study participants will also be invited to complete the baseline questionnaire.

Length of study:

* The LS tumor screening portion of the OCCPI will take 1-4 months.
* If applicable, genetic testing results should be ready in an additional 3-6 months.
* Overall, your participation in the LS screening portion of the OCCPI is expected to take about 1 year. Most of this time will be spent waiting for results. Your active involvement will take about 15 minutes on the day that you provide consent and about 60 minutes when you complete the questionnaire from home.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with colorectal adenocarcinoma (all stages) and have a resection at any hospital in Ohio between 1/1/2013 and 12/31/2016.

   * For individuals who have neoadjuvant treatment and show a complete response at resection, the tumor screening will be attempted on their original biopsy (even if it occurred in 2012) as long as their resection occurred between 1/1/2013 and 12/31/2016.
   * Many individuals with stage IV CRC will not have a resection; therefore, the tumor screening will be attempted on their original colon biopsy as long as their primary diagnosis occurred between 1/1/2013 and 12/31/2016. If only metastatic CRC is available on a biopsy (liver or lymph node metastases), tumor screening will be attempted on the metastatic tissue.
2. Newly diagnosed with endometrial cancer (any histology except sarcoma) and have a resection between 1/1/2013 and 12/31/2016 at OSU only.
3. All at-risk relatives of the participants found to have LS.
4. First-degree relatives (parents, siblings and adult children ≥ 25 years of age) of the CRC participants who do not have LS.

Exclusion Criteria:

1. Prisoners.
2. Individuals who are under the age of 18.
3. Individuals must have a primary colorectal or endometrial cancer, not a recurrence of a previous colorectal or endometrial cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3470 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Determine the Incidence of Hereditary Cancer Syndromes among Newly Diagnosed Colorectal Cancer Patients | 36 months (initial assessment)
  Through tumor testing for Lynch syndrome and follow-up genetic testing for all patients with abnormal tumor testing and select patients with normal tumor testing (those diagnosed under age 50 and those at or over age 50 with a first degree relative with colorectal or endometrial cancer or synchronous or metachronous colon or endometrial cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hampel, MS, LGC, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (49):
- United States (49):
  - Akron General Medical Center, Akron, Ohio
  - Akron City/St. Thomas Hospital (Summa Health System), Akron, Ohio
  - Summa Barberton (Summa Health System), Barberton, Ohio
  - Mercy Clermont, Batavia, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Hospital, Canton, Ohio
  - Adena Health System, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital (TriHealth), Cincinnati, Ohio
  - Bethesda North Hospital (TriHealth), Cincinnati, Ohio
  - Mercy Anderson, Cincinnati, Ohio
  - Mercy West, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - MetroHealth, Cleveland, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Summa Western Reserve (Summa Health System), Cuyahoga Falls, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Good Samaritan Hospital Dayton, Dayton, Ohio
  - Kettering Medical Center, Dayton, Ohio
  - Wright-Patterson Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Fairfield, Fairfield, Ohio
  - Blanchard Valley Health System, Findlay, Ohio
  - Wayne Healthcare, Greenville, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Marion General Hospital, Marion, Ohio
  - St. Luke's Hospital (ProMedica), Maumee, Ohio
  - Toledo Clinic Cancer Center, Maumee, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Atrium Medical Center, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Robinson Memorial (Summa Health System), Ravenna, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital (ProMedica Health System), Sylvania, Ohio
  - Toledo Hospital (Promedica Health System), Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Genesis Cancer Care Center (Genesis Healthcare System), Zanesville, Ohio

REFERENCES:
- [Background] Hampel H, Frankel WL, Martin E, Arnold M, Khanduja K, Kuebler P, Nakagawa H, Sotamaa K, Prior TW, Westman J, Panescu J, Fix D, Lockman J, Comeras I, de la Chapelle A. Screening for the Lynch syndrome (hereditary nonpolyposis colorectal cancer). N Engl J Med. 2005 May 5;352(18):1851-60. doi: 10.1056/NEJMoa043146. PMID 15872200
- [Background] Hampel H, Frankel WL, Martin E, Arnold M, Khanduja K, Kuebler P, Clendenning M, Sotamaa K, Prior T, Westman JA, Panescu J, Fix D, Lockman J, LaJeunesse J, Comeras I, de la Chapelle A. Feasibility of screening for Lynch syndrome among patients with colorectal cancer. J Clin Oncol. 2008 Dec 10;26(35):5783-8. doi: 10.1200/JCO.2008.17.5950. Epub 2008 Sep 22. PMID 18809606
- [Background] Palomaki GE, McClain MR, Melillo S, Hampel HL, Thibodeau SN. EGAPP supplementary evidence review: DNA testing strategies aimed at reducing morbidity and mortality from Lynch syndrome. Genet Med. 2009 Jan;11(1):42-65. doi: 10.1097/GIM.0b013e31818fa2db. No abstract available. PMID 19125127
- [Background] Evaluation of Genomic Applications in Practice and Prevention (EGAPP) Working Group. Recommendations from the EGAPP Working Group: genetic testing strategies in newly diagnosed individuals with colorectal cancer aimed at reducing morbidity and mortality from Lynch syndrome in relatives. Genet Med. 2009 Jan;11(1):35-41. doi: 10.1097/GIM.0b013e31818fa2ff. PMID 19125126
- See also: The Jamesline — http://cancer.osu.edu